CLINICAL TRIAL: NCT04612478
Title: Use of a Self-Directed Exercise Program (SDEP) Following Selected Lower Extremity Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00082966; Pro00024283 (Other: Atrium)
Record Dates: First submitted 2018-05-07; First posted 2020-11-03 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Musculoskeletal Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinic-Based Physical Therapy (Other): Patients will be referred to PT by the orthopaedic surgeon for enrollment into a clinic-based PT program per usual referral patterns at the surgeon's center. Patients will receive services based on their health care benefits defined by his or her insurance plan.
  Interventions: Behavioral: Clinic-Based Physical
- Self-Directed Exercise Program (Other): The full SDEP program, which will be developed by physical therapists, orthopaedic trauma surgeons, and investigators with experience in health behavior change, will be designed to maximize adherence/compliance with the program. The SDEP manual will provide detailed instructions on exercises, such as repetitions, frequency, and required equipment, which can be implemented in the home environment. The basis for the exercise regimen is derived from the American Academy of Orthopaedic Surgeons (AAOS) sample home based exercise program available in handout form. The program provides instructions on exercises, repetitions or duration, frequency, and required equipment which can be implemented in the home environment.
  Interventions: Behavioral: Self-Directed Exercise Program
- Observational (No Intervention): Patients who are unwilling to be randomized will be enrolled in an observational arm of the study. They will be asked to complete all baseline and follow-up assessments, and participation in formal PT or SDEP will be documented.

INTERVENTIONS:
Behavioral: Self-Directed Exercise Program — The full SDEP program, which will be developed by physical therapists, orthopaedic trauma surgeons, and investigators with experience in health behavior change, will be designed to maximize adherence/compliance with the program
  Arms: Self-Directed Exercise Program
Behavioral: Clinic-Based Physical — Patients will be referred to PT by the orthopaedic surgeon for enrollment into a clinic-based PT program per usual referral patterns at the surgeon's center. Patients will receive services based on their health care benefits defined by his or her insurance plan.
  Arms: Clinic-Based Physical Therapy

SUMMARY:
The purpose of this study is to compare the effectiveness and value of clinic-based physical therapy (PT) and a home-based, self-directed exercise program (SDEP). The home exercise program will be developed by a team of physical therapists, orthopaedic trauma surgeons and experts in rehabilitation engagement in collaboration with patients recovering from traumatic lower-extremity injuries. The study will also determine which subgroups of individuals based on patient and injury characteristics are the best candidates for a home exercise program.

DETAILED DESCRIPTION:
There is little clinical debate that patients with multiple extremity injuries or injuries with associated complex soft tissue damage or nerve deficits benefit from supervised PT. Prior research from the LEAP Study examined the impact of PT on patients with high energy trauma injuries below the distal femur.1 While the surgeons and PTs differed in their assessment of perceived need for PT,2,3 evidence demonstrates the beneficial effect of PT for this patient population.4 Research on combat-related lower extremity limb salvage patients showed a significant benefit and a higher return-to-duty rate following intense and focused rehabilitation combined with an integrated orthotic.5-7 However, the majority of lower extremity fractures seen in the military and civilian sectors are not combat related or of the severity of the Lower Extremity Assessment Project (LEAP) limb salvage patients and, thus may not require intensive, clinic-based, supervised PT treatment. Patients with isolated major lower extremity fractures may benefit from a self-guided, home-based post-injury exercise program. Studies evaluating home exercise programs for elective orthopaedic reconstruction surgery for joint replacement and anterior cruciate ligament (ACL )reconstruction have reported equivalent outcomes compared to in-person, supervised PT.8-12 Because PT resources are critical, limited, and expensive in most civilian centers, identifying the patients who would most benefit from utilizing these resources could result in savings for both the patients and the health care systems, and lead to more efficient access to PT services by the population who needs them the most. In addition to health systems benefits, patients able to achieve positive outcomes through a home-based, self-directed exercise program would experience flexibility regarding when the exercises are performed.

The purpose of this study is to compare the effectiveness and value of clinic-based PT and a home-based, self-directed exercise program (SDEP). The home exercise program will be developed by a team of physical therapists, orthopaedic trauma surgeons and experts in rehabilitation engagement in collaboration with patients recovering from traumatic lower-extremity injuries. The study will also determine which subgroups of individuals based on patient and injury characteristics are the best candidates for a home exercise program.

Hypothesis: The overall hypothesis is that return to work/major activities as well as clinical and functional outcomes and health-related quality of life for patients who receive clinic-based PT will be similar to patients receiving SDEP.

Specific Aim 1: To compare the effectiveness of SDEP, exercise instructions given by physician and clinic-based PT for improving return to work/major activities, clinical and functional/performance outcomes and health-related quality of life in patients following selected lower-extremity fractures.

Specific Aim 2: To determine which sub-groups of patients, based on patient and injury characteristics, are most likely to benefit from SDEP.

Specific Aim 3: To compare the cost-effectiveness of clinic-based PT and SDEP

.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 with operative fractures of the femur and tibia (to include distal femur (33A, B), plateau (41A, B), pilon (43A, B), and selected ankle injuries (44A, B)) presenting to the Orthopaedic Surgeon for either acute care or for the follow-up of care performed elsewhere (within 14 days of the injury).
* All patients must be English or Spanish competent and able to be followed at the sites for at least 12 months following injury.

Exclusion Criteria:

* Patients with Injury Severity Score (ISS)>18
* Bilateral lower-extremity injuries that preclude crutch ambulation
* Associated spine, pelvic, and/or acetabular fractures that otherwise alter weightbearing plan
* Type III B/C open fractures
* Glasgow Coma Scale <15 at time of discharge
* Major peripheral nerve injury
* Planned admission to a skilled nursing facility or inpatient rehabilitation facility
* Pregnant women
* Patients diagnosed with a Traumatic Brain Injury (TBI) will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Return to work/major activities | 12 months
  Measured through the rate of return to work/duty 12 months post discharge using the Work Productivity and Activity Impairment Questionnaire (WPAI)

SECONDARY OUTCOMES:
Change in Quality of Life | baseline, 3, 6 and12 months
  The PROMIS-29 Profile v2.0 assesses depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities. Raw scores range from 4-20, with higher scores indicating lower quality of life in that area, except for the sleep disturbance sub-section, where higher scores indicate better sleep.
Kinesiophobia | baseline, 3, 6 and12 months
  As measured by Tampa Scale for Kinesiophobia (TSK). The TSK is a self-completed questionnaire and the range of scores are from 17 to 68 where the higher scores indicate an increasing degree of kinesiophobia
Time to Radiographic Fracture Healing | 3, 6 & 12 months
  Radiographs will be assessed for fracture healing.
Muscle Strength | 12 months
  Muscle strength will be measured using a dynamometer.
Joint Range of Motion (ROM) | 12 months
  Joint range of motion will be measured using a goniomenter.
Resilience | Baseline, 3, 6 & 12 months
  Resiliency will be measured using the Connor-Davidson Resilience Scale. Total Score of the resilience questions is 0 to 40, 10 subscales from 0 to 4 (summed up for total score), the higher the score the better the resilience

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Seymour, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Carolinas Medical Center, Charlotte, North Carolina
  - Greenville Health System, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bosse MJ, MacKenzie EJ, Kellam JF, Burgess AR, Webb LX, Swiontkowski MF, Sanders RW, Jones AL, McAndrew MP, Patterson BM, McCarthy ML, Travison TG, Castillo RC. An analysis of outcomes of reconstruction or amputation after leg-threatening injuries. N Engl J Med. 2002 Dec 12;347(24):1924-31. doi: 10.1056/NEJMoa012604. PMID 12477942
- [Background] Castillo RC, MacKenzie EJ, Webb LX, Bosse MJ, Avery J; LEAP Study Group. Use and perceived need of physical therapy following severe lower-extremity trauma. Arch Phys Med Rehabil. 2005 Sep;86(9):1722-8. doi: 10.1016/j.apmr.2005.03.005. PMID 16181933
- [Background] Archer KR, Mackenzie EJ, Castillo RC, Bosse MJ; LEAP Study Group. Orthopedic surgeons and physical therapists differ in assessment of need for physical therapy after traumatic lower-extremity injury. Phys Ther. 2009 Dec;89(12):1337-49. doi: 10.2522/ptj.20080200. Epub 2009 Oct 29. PMID 19875460
- [Background] Castillo RC, MacKenzie EJ, Archer KR, Bosse MJ, Webb LX; LEAP Study Group. Evidence of beneficial effect of physical therapy after lower-extremity trauma. Arch Phys Med Rehabil. 2008 Oct;89(10):1873-9. doi: 10.1016/j.apmr.2008.01.032. PMID 18929015
- [Background] Blair JA, Patzkowski JC, Blanck RV, Owens JG, Hsu JR; Skeletal Trauma Research Consortium (STReC). Return to duty after integrated orthotic and rehabilitation initiative. J Orthop Trauma. 2014 Apr;28(4):e70-4. doi: 10.1097/BOT.0000000000000006. PMID 24121984
- [Background] Bedigrew KM, Patzkowski JC, Wilken JM, Owens JG, Blanck RV, Stinner DJ, Kirk KL, Hsu JR; Skeletal Trauma Research Consortium (STReC). Can an integrated orthotic and rehabilitation program decrease pain and improve function after lower extremity trauma? Clin Orthop Relat Res. 2014 Oct;472(10):3017-25. doi: 10.1007/s11999-014-3609-7. PMID 24744130
- [Background] Patzkowski JC, Owens JG, Blanck RV, Kirk KL, Hsu JR; Skeletal Trauma Research Consortium (STReC). Deployment after limb salvage for high-energy lower-extremity trauma. J Trauma Acute Care Surg. 2012 Aug;73(2 Suppl 1):S112-5. doi: 10.1097/TA.0b013e3182606291. PMID 22847079
- [Background] Moffet H, Tousignant M, Nadeau S, Merette C, Boissy P, Corriveau H, Marquis F, Cabana F, Ranger P, Belzile EL, Dimentberg R. In-Home Telerehabilitation Compared with Face-to-Face Rehabilitation After Total Knee Arthroplasty: A Noninferiority Randomized Controlled Trial. J Bone Joint Surg Am. 2015 Jul 15;97(14):1129-41. doi: 10.2106/JBJS.N.01066. PMID 26178888
- [Background] Fischer DA, Tewes DP, Boyd JL, Smith JP, Quick DC. Home based rehabilitation for anterior cruciate ligament reconstruction. Clin Orthop Relat Res. 1998 Feb;(347):194-9. PMID 9520889
- [Background] Grant JA, Mohtadi NG. Two- to 4-year follow-up to a comparison of home versus physical therapy-supervised rehabilitation programs after anterior cruciate ligament reconstruction. Am J Sports Med. 2010 Jul;38(7):1389-94. doi: 10.1177/0363546509359763. Epub 2010 Apr 1. PMID 20360607
- [Background] Grant JA, Mohtadi NG, Maitland ME, Zernicke RF. Comparison of home versus physical therapy-supervised rehabilitation programs after anterior cruciate ligament reconstruction: a randomized clinical trial. Am J Sports Med. 2005 Sep;33(9):1288-97. doi: 10.1177/0363546504273051. Epub 2005 Jul 7. PMID 16002493
- [Background] Ferguson C, Harmer L, Seymour RB, Ellington K, Bosse MJ, and the CMC-OC Ankle Fracture Study Group. Does Physical Therapy Predict Outcomes after Ankle Fractures and Ankle Fracture-Dislocations? Podium Presentation, Orthopaedic Trauma Association Annual Meeting, October 2015.
- [Background] Darter BJ, Nielsen DH, Yack HJ, Janz KF. Home-based treadmill training to improve gait performance in persons with a chronic transfemoral amputation. Arch Phys Med Rehabil. 2013 Dec;94(12):2440-2447. doi: 10.1016/j.apmr.2013.08.001. Epub 2013 Aug 13. PMID 23954560
- [Background] Ravaud P, Giraudeau B, Logeart I, Larguier JS, Rolland D, Treves R, Euller-Ziegler L, Bannwarth B, Dougados M. Management of osteoarthritis (OA) with an unsupervised home based exercise programme and/or patient administered assessment tools. A cluster randomised controlled trial with a 2x2 factorial design. Ann Rheum Dis. 2004 Jun;63(6):703-8. doi: 10.1136/ard.2003.009803. PMID 15140778
- [Background] Lim HJ, Moon YI, Lee MS. Effects of home-based daily exercise therapy on joint mobility, daily activity, pain, and depression in patients with ankylosing spondylitis. Rheumatol Int. 2005 Apr;25(3):225-9. doi: 10.1007/s00296-004-0536-z. Epub 2005 Jan 14. PMID 15650833
- [Background] Shirado O, Doi T, Akai M, Hoshino Y, Fujino K, Hayashi K, Marui E, Iwaya T; Japan Low back-pain Exercise Therapy Study; Investigators Japanese Orthopaedic Association; Japanese Society for Musculoskeletal Rehabilitation; Japanese Clinical Orthopaedic Association. Multicenter randomized controlled trial to evaluate the effect of home-based exercise on patients with chronic low back pain: the Japan low back pain exercise therapy study. Spine (Phila Pa 1976). 2010 Aug 1;35(17):E811-9. doi: 10.1097/BRS.0b013e3181d7a4d2. PMID 20628332
- [Background] Valdes K, Naughton N, Burke CJ. Therapist-supervised hand therapy versus home therapy with therapist instruction following distal radius fracture. J Hand Surg Am. 2015 Jun;40(6):1110-6.e1. doi: 10.1016/j.jhsa.2015.01.036. Epub 2015 Mar 25. PMID 25817323
- [Background] Souer JS, Buijze G, Ring D. A prospective randomized controlled trial comparing occupational therapy with independent exercises after volar plate fixation of a fracture of the distal part of the radius. J Bone Joint Surg Am. 2011 Oct 5;93(19):1761-6. doi: 10.2106/JBJS.J.01452. PMID 22005860
- [Background] Gleyze P, Georges T, Flurin PH, Laprelle E, Katz D, Clavert P, Charousset C, Levigne C; French Arthroscopy Society. Comparison and critical evaluation of rehabilitation and home-based exercises for treating shoulder stiffness: prospective, multicenter study with 148 cases. Orthop Traumatol Surg Res. 2011 Dec;97(8 Suppl):S182-94. doi: 10.1016/j.otsr.2011.09.005. Epub 2011 Oct 28. PMID 22036242
- [Background] Schrader J, Tebbe U, Borries M, Ruschitzka F, Schoel G, Kandt M, Warneke G, Zuchner C, Weber MH, Neu U, et al. [Plasma endothelin in normal probands and patients with nephrologic-rheumatologic and cardiovascular diseases]. Klin Wochenschr. 1990 Aug 2;68(15):774-9. doi: 10.1007/BF01647248. German. PMID 2214602
- [Background] Hayes K, Ginn KA, Walton JR, Szomor ZL, Murrell GA. A randomised clinical trial evaluating the efficacy of physiotherapy after rotator cuff repair. Aust J Physiother. 2004;50(2):77-83. doi: 10.1016/s0004-9514(14)60099-4. PMID 15151491
- [Background] Hohmann E, Tetsworth K, Bryant A. Physiotherapy-guided versus home-based, unsupervised rehabilitation in isolated anterior cruciate injuries following surgical reconstruction. Knee Surg Sports Traumatol Arthrosc. 2011 Jul;19(7):1158-67. doi: 10.1007/s00167-010-1386-8. Epub 2011 Jan 26. PMID 21267543
- [Background] Swiontkowski MF, Engelberg R, Martin DP, Agel J. Short musculoskeletal function assessment questionnaire: validity, reliability, and responsiveness. J Bone Joint Surg Am. 1999 Sep;81(9):1245-60. doi: 10.2106/00004623-199909000-00006. PMID 10505521
- [Background] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT04612478/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT04612478/ICF_001.pdf